CLINICAL TRIAL: NCT02812667
Title: A Phase I Study of Nivolumab in Combination With Escalating Doses of Plinabulin in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Nivolumab in Combination With Plinabulin in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lyudmila Bazhenova, M.D. (Other)
Collaborators: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lyudmila Bazhenova, M.D., Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160186
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Metastatic; NSCLC; nivolumab; plinabulin; BPI-2358; opdivo; Non-Small Cell Lung Cancer; cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Nivolumab; NPI 2358

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab + Plinabulin (Experimental): Nivolumab 240mg IV, day 1 and 15 until disease progression Plinabulin 3.5mg/m2, 20mg/m2, 30 mg/m2 or 40mg/m2 IV, day 1,8 and 15 until disease progression
  Interventions: Drug: Nivolumab + Plinabulin

INTERVENTIONS:
Drug: Nivolumab + Plinabulin

SUMMARY:
The purpose of the study is to determine whether plinabulin (also known as BPI-2358) has an effect on cancer and body in combination with nivolumab, a standard treatment for metastatic squamous non-small cell lung cancer with progression on or after platinum-based chemotherapy.

Plinabulin inhibits tumor growth by targeting both new and existing blood vessels going to the tumor as well as killing tumor cells. Plinabulin is an investigational drug, a drug that is not approved for use outside of research studies by regulatory agencies. Up to 38 patients will be enrolled.

DETAILED DESCRIPTION:
Plinabulin is a microtubule destabilizing agent (MDA) that inhibits the polymerization of tubulin monomers with resultant vascular disrupting properties. Plinabulin inhibits tumor growth by targeting both angiogenesis and tumor vasculature as well as directly by inducing apoptosis via the Ras-JNK pathway. It also may activate anti-tumor immunity via inducing maturation of dendritic cells (DC) and triggering release of pro-inflammatory cytokines. Plinabulin could therefore have a synergic anti-tumor effect when combined with immune-checkpoint inhibitors. This hypothesis has been confirmed in a murine model bearing subcutaneous MC38 colon cancers using other MDAs, including ansamitocin P3, which induces DC maturation similar to that of plinabulin. Plinabulin has been tested in a randomized phase 2 trial in combination of docetaxel and showed similar response rate to that of docetaxel alone, but with a significantly longer duration of response.

Nivolumab is an inhibitor of the programmed cell death receptor-1 checkpoint pathway (PD-1) that has superior activity in NSCLC, regardless of tumor histology, comparing to standard of care. In this study, we plan to combine nivolumab with escalating doses of plinabulin to determine the maximum tolerated dose (MTD) and /or recommended Phase 2 dose (RP2D) of the combination. An expansion cohort will be enrolled at RP2D to further assess toxicities and to evaluate preliminary anti-tumor activity.

This is a single-center, phase 1 dose finding trial of plinabulin, combining with FDA approved dose of nivolumab, using a 3+3 design in patients with metastatic NSCLC who progressed after chemotherapy, including a platinum-containing regimen. Patients will receive plinabulin at escalating doses in combination with nivolumab. Doses of plinabulin and nivolumab will be administered as intravenous infusions in 4-week cycles. Patients will receive both medications on Days 1 and 15 and additional dose of plinabulin on Day 8. Plinabulin will be administered 60 minutes after the completion of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically-confirmed metastatic NSCLC whose disease progressed during/after treatment with at least one platinum-containing chemotherapy regimen.
* At least 1 prior systemic therapy for metastatic disease. Adjuvant chemotherapy or concurrent chemoradiation for early stage disease does not count as prior therapy unless patients progressed within 6 months of completion of chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
* Life expectancy ≥ 12 weeks
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST).
* Adequate hematopoietic, electrolyte, hepatic, and renal laboratory findings.
* Prior chemotherapy must have been completed at least 4 weeks or at least 5 half-lives (whichever is longer) before study drug administration, and all adverse events have either returned to baseline or stabilized
* Prior treated brain metastases are allowed. However, prior treated brain metastases must be without MRI evidence of progression for at least 4 weeks and off systemic steroids for at least 2 weeks before study drug administration
* Prior definitive radiation therapy must have been completed at least 4 weeks before study drug administration. Prior palliative radiotherapy should be completed at least 2 weeks before study drug administration. Whole brain radiation therapy (WBRT), stereotactic radiosurgery (SRS) and focal radiation to the sites of pain or bronchial obstruction will be considered palliative. No radiopharmaceuticals (strontium, samarium) within 8 weeks before study drug administration
* Prior major surgery must be completed at least 4 weeks before study drug administration. Prior minor surgery must be completed at least 1 week before study drug administration and subjects should be recovered. Percutaneous biopsies should be completed at least 10 days prior to study drug administration;
* A negative serum pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

* History of grade 3 or above hypersensitivity reactions to other monoclonal antibodies
* Subjects with a history of a cardiovascular illness.
* Uncontrolled hypertension, SBP> 160 or DBP>100
* Symptomatic or untreated brain metastases
* Presence of leptomeningeal disease
* Pulmonary conditions, which in the PI's opinion would increase the risk of immunotherapy-related pulmonary toxicity.
* Has active, non-infectious pneumonitis
* Presence of a second malignancy, excluding non-melanomatous skin cancer unless in remission for 3 years
* Subjects with any active, known, or suspected autoimmune disease.
* History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
* Prior therapy with microtubule destabilizing agents for NSCLC (ie. Vinorelbine)
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-stimulation pathways);
* Known history of Human Immunodeficiency Virus;
* Active infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA)
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events
* Concurrent medical condition requiring the use of immunosuppressive medications, or systemic steroids.
* Use of other investigational drugs within 28 days or at least 5 half-lives before study drug administration
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years
Frequency and severity of treatment-related adverse events as assessed by CTCAE v4. | 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
Disease control rate (DCR) | 2 years
Progression free survival (PFS) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lyudmilla Bazhenova, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States